CLINICAL TRIAL: NCT03438149
Title: Microparticles as a Biomarker of Incident Cardiovascular Risk in Patients With Obstructive Sleep Apnea
Brief Title: Microparticles in Obstructive Sleep Apnea
Acronym: BioSAS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-A02494-49
Record Dates: First submitted 2018-02-02; First posted 2018-02-19 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Sleep Apnea, Obstructive
Keywords: microparticles; cardiovascular outcomes
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Obstructive sleep apnea (OSA) is independently associated with cardiovascular diseases, including myocardial infarction and stroke. OSA may promote atherosclerosis risk factors such as hypertension, diabetes and dyslipidemia and may have direct proatherogenic effects on the vascular wall. A growing number of studies have recently focused on the role of microparticles (MPs) in the atherogenic process. Case-control studies have shown that platelet-, endothelial- and leukocyte-derived MP levels are increased in OSA and that leukocyte-derived MP are released during the night in OSA. Furthermore, experimental evidence shows that MPs from OSA patients induce endothelial dysfunction.

The objective of this prospective study is to evaluate the impact of increased levels of leukocyte derived MPs on the cardiovascular outcomes in patients with prevalent cardiovascular diseases investigated for OSA.

DETAILED DESCRIPTION:
MPs are small plasma membrane vesicles that can be released by a variety of vascular or blood cells and that contain membrane and cytosolic elements. Case-control studies have shown that platelet-, endothelial- and leukocyte-derived MP levels are increased in OSA. Experimental evidence shows that MPs from OSA patients induce endothelial dysfunction, inflammation, and vascular hyperreactivity when injected to mice.

The impact of increased levels of MPs on the cardiovascular prognosis in OSA patient with prevalent cardiovascular diseases in unknown.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of coronary artery disease or cerebrovascular disease
* diagnosis of moderate-to-severe OSA

Exclusion Criteria:

* pregnancy
* previously treated OSA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with prevalent cardiovascular diseases referred to a sleep clinic for suspected OSA.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
death from any cardiovascular cause | first event within 5 years after inclusion
  outcomes assessed every year at the follow up visit or by calling the primary care physician
myocardial infarction (acute infarct or silent myocardial infarction or unstable angina) | first event within 5 years after inclusion
  outcomes assessed every year at the follow up visit or by calling the primary care physician
cerebrovascular infarction (stroke or transient ischemic attack) | first event within 5 years after inclusion
  outcomes assessed every year at the follow up visit or by calling the primary care physician
hospitalization for heart failure | first event within 5 years after inclusion
  outcomes assessed every year at the follow up visit or by calling the primary care physician

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratoire du Sommeil, Département de Pneumologie, CHU d'Angers, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided